CLINICAL TRIAL: NCT04842331
Title: A Randomised Multicentre Post-exposure Prophylaxis Clinical Trial Evaluating RESP301, an Inhaled Therapy for Treatment of Lung Infections, for Prevention of Onward Transmission of Viral Infections Including SARS-CoV-2 to Household Members
Brief Title: PREvent Viral Exposure and Transmission Study: a COVID-19 (SARS-CoV-2) PEP Study (PREVENT)
Acronym: PREVENT
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: A combination of factors, including the dynamic nature of the COVID-19 pandemic and the successful vaccination program, has resulted in a very sharp decline in the number of patients with COVID-19
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RESP301-006
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Viral Infection; Respiratory Tract Diseases; COVID-19 Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients are randomised to 1 of 2 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RESP301 + Standard of Care (SOC) (Experimental): Treatment arm will receive the study drug RESP301 alongside standard of care (SOC).
  RESP301 will be administered for a period of 7 days (i.e. 21 doses) to both index cases and their household members in the treatment arm. Participants will be given the first dose under medical supervision and self-administer at home the remaining 20 doses.
  RESP301 is a formulation consisting of 3 agents currently used in clinical practice: mannitol, sodium nitrite and citric acid.
  Interventions: Drug: RESP301 (a nitric oxide generating solution); Drug: Standard of Care (SOC)
- Standard of Care (SOC) (Active Comparator): SOC
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: RESP301 (a nitric oxide generating solution) — Administration is simple and convenient; each dose of RESP301 is administered 3 times daily (at least 4 hours apart) via inhalation using a portable handheld vibrating mesh nebuliser for approximately 8-10 minutes.
  Arms: RESP301 + Standard of Care (SOC)
Drug: Standard of Care (SOC) — Participants will receive institutional SOC for the treatment.

SUMMARY:
This is an open label controlled household-randomised trial designed to evaluate the efficacy of RESP301 alongside standard of care ("SOC") versus SOC alone.

DETAILED DESCRIPTION:
In this study, RESP301 is investigated as a post-exposure prophylaxis (PEP). RESP301 is a liquid which is inhaled using a handheld nebuliser and produces Nitric Oxide, which is also naturally produced in the human body and is a key part of our defence against infections in the lungs. In a laboratory setting,RESP301 has been shown to be highly effective against many respiratory viruses, including CoV2 and influenza.

RESP301 is currently being used as treatment for hospitalised COVID-19 patients in an ongoing clinical trial.

The aim of this PEP study is to prevent onward transmission of the infection within households by treating both the infected individual and their household members. The primary endpoint is to evaluate the incidence of newly confirmed CoV2 infection (PCR positive) in previously uninfected household members (PCR negative, antibody negative and unvaccinated) of CoV-2 positive index cases after a 7 day course of treatment.

Participants who are not eligible to participate, or do not want to participate will be invited to take part in an optional study where the participants will be asked to complete a short questionnaire.

Participants will be on the study for a total duration of 15-17 days. Approximately 600 adults will be on the study in total and index cases will be randomised 1:1 to either RESP301 (plus SOC) or SOC alone, with all eligible persons in the same household enrolled into the same treatment arm.

The study will be divided into the following periods: Baseline Visit / screening (1 day): Treatment Period (self administered at home - 7 days): End of Treatment Period (1 day): Follow-Up Period (~5-7 days): Follow-Up Call (1 day between day 15-17)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Able to give written informed consent
3. Index cases: presenting with mild/moderate viral infection symptoms, who the Investigator considers can be treated at home.
4. Negative pregnancy test for women of childbearing age at Baseline visit (includes screening).
5. Able to operate and maintain nebuliser, as assessed by the Investigator.

Exclusion Criteria:

1. Both Index cases and Household members: Unable to tolerate use of a nebuliser for approximately 8-10 minutes as required by the study according to Investigator's opinion
2. Both Index and Household members:

   1. Any unstable, uncontrolled or severe medical condition which in the opinion of the investigator would make the participant unsuitable for the trial
   2. COPD/Asthma or any severe respiratory disease requiring the use of oral steroids or biologics
3. Participation in other clinical investigations utilising investigational treatment within the last 30 days / 5 half-lives whichever is longer
4. Participant lives at home with no other potentially eligible adults in the household
5. Women of childbearing age unable or unwilling to use an adequate form of contraception for the duration of the study i.e. double barrier contraceptives.
6. Male participants who are unwilling or unable to use an effective method of contraception for the duration of the study.
7. Known allergy/hypersensitivity to or relevant drug-drug interaction with study drug/components of study drug
8. History of methaemoglobinaemia
9. Deemed unlikely to be able to adhere to protocol in view of investigator
10. Any subject who in the opinion of the investigator would not be best served by participating in this clinical trial
11. Prescribed Nitric Oxide donating agents (e.g. Nitroprusside, Isosorbide dinitrate, Isosorbide mononitrate, Naproxcinod, Molsidomine and Linsidomine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
PCR positive and negative | Day 1-7
  PCR positive cases in previously uninfected household members (PCR negative, antibody negative and unvaccinated) of CoV-2 positive index cases after a 7 day course of treatment.

SECONDARY OUTCOMES:
Percentage (%) of participants able to tolerate the test dose | Day 1
  Percentage (%) of participants able to tolerate the test dose, i.e. without any treatment-related AE at the Baseline Visit that led to participant not being able to continue with the remaining doses
Percentage (%) of total doses taken | Day 1-7
  Compliance with RESP301 administration schedule by enrolled participants over the treatment period (% of total doses taken).

CONTACTS AND LOCATIONS:
Overall Officials: Onn Min Kon, Professor, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom